CLINICAL TRIAL: NCT05807685
Title: The Effect Of Laughter Therapy On Burnout And Guılt In Women Wıth Chıldren In Prımary School
Brief Title: The Effect Of Laughter Therapy On Burnout And Guılt In Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: sinopUberna-1
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Laughter; Burnout
Keywords: laughter therapy; burnout; guilt; women
MeSH Terms: conditions — Laughter; Burnout, Psychological | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): At the beginning of the study, Data collection tools such as Individual Identification Form, Expressed Guilt Scale and Burnout Scale Short Version will be applied to the control group.
  No intervention will be made in the control group. In the post-test, the Expressed Guilt Scale and the Burnout Scale Short Version will be administered again.
- experimental group (Experimental): Arm Title: Experimental Group: Individual Identification Form, Expressed Guilt Scale and Burnout Scale Short Version will be administered to the mothers of children studying at Sinop Atatürk Primary School in the 2022-2023 spring semester before the laughter therapy. At the end of the laughter therapy, the Expressed Guilt Scale and the Short Version of the Burnout Scale will be administered as a post-test.
  The Individual Identification Form, Expressed Guilt Scale and Burnout Scale Short Version will be used for all mothers of the students studying in Atatürk Primary School in the 2022-2023 academic year. All women whose Burnout Scale Short Form is above the average will be included in the study. Since all women whose Burnout Scale Short Form is above the average, who volunteered to participate in the study and who met the inclusion criteria will be included in the study, no additional sample selection will be made.
  Interventions: Behavioral: laughter therapy

INTERVENTIONS:
Behavioral: laughter therapy — Description: Laughter therapy session will be applied online for 25-30 minutes once a week for 2 months by the researchers who has the Laughter therapy certificate to the application group. In the laughter therapy session, the practices of introducing the practitioner and introducing the therapy, breathing exercises for a healthy life, keeping the rhythm accompanied by music, turning the laughter that started as if it were childlike games into reality will be carried out.
  Arms: experimental group

SUMMARY:
: Responsibility of women staying in their traditional and modern roles has increased and the difficulties experienced by women require them to struggle with many problems. As a result of these experiences, problems have arisen for women. In addition to the intensity of the home/work life of women who have children in primary school, the lesson and responsibility of the child falls on the women. In a patriarchal society, burdening all non-working women with the responsibility of their child in addition to housework increases the fatigue of mothers. Due to this intensity, they are not able to spare time for themselves and feel guilty. In women, this situation gradually causes burnout syndrome. One of the most important personal development methods used to reduce burnout is laughter therapy. The aim of this study is to apply laughter therapy in order to reduce this sense of burnout and guilt in women.

Aim: In this study, it was aimed to examine the effect of laughter therapy on the feelings of burnout and guilt of women who have children at primary school age.

DETAILED DESCRIPTION:
Detailed Description: Method: The research is a randomized controlled experimental study.

The research will be carried out with the mothers of the students studying at Sinop Atatürk Primary School in the 2022-2023 academic year.

Research Population and Sample: All of the mothers of the students studying at the determined Sinop Atatürk Primary School in the spring term of 2022-2023 will form the universe. The sample of the study will include all mothers of the students studying at Sinop Atatürk Primary School in the 2022-2023 academic spring term, who meet the inclusion criteria, have a burnout scale score of 3.5 and above, and volunteer to participate in the research.

Arm Title: Control Group: At the beginning of the study, Data collection tools such as Individual Identification Form, Expressed Guilt Scale and Burnout Scale Short Version will be applied to the control group.

No intervention will be made in the control group. In the post-test, the Expressed Guilt Scale and the Burnout Scale Short Version will be administered again.

Arm Title: Experimental Group: Individual Identification Form, Expressed Guilt Scale and Burnout Scale Short Version will be administered to the mothers of children studying at Sinop Atatürk Primary School in the 2022-2023 spring semester before the laughter therapy. At the end of the laughter therapy, the Expressed Guilt Scale and the Short Version of the Burnout Scale will be administered as a post-test.

The Individual Identification Form, Expressed Guilt Scale and Burnout Scale Short Version will be used for all mothers of the students studying in Atatürk Primary School in the 2022-2023 academic year. All women whose Burnout Scale Short Form is above the average will be included in the study. Since all women whose Burnout Scale Short Form is above the average, who volunteered to participate in the study and who met the inclusion criteria will be included in the study, no additional sample selection will be made. The application and control group will be determined on random.org among the group that constitutes the sample of the study. A 30-minute laughter therapy session will be applied to the application group once a week for 2 months. At the end of two months, the Expressed Guilt Scale and the Short Version of the Burnout Scale will be administered to both the application group and the control group.

ELIGIBILITY:
Inclusion Criteria:

Being the mother of the child studying at Sinop Atatürk Primary School where the research will be conducted, Having a burnout scale score of 3.5 and above, Volunteer to participate in research.

Exclusion Criteria:

Not having a child studying at the Sinop Atatürk Primary School where the research will be conducted, Being the father of the child who was educated at the Sinop Atatürk Primary School, where the research will be conducted, Having a burnout scale score below 3.5, Not volunteering to participate in the research.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-10 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Expressed Guilt Scale | one day
  The scale developed by Guerrero et al. (2009) consists of 20 items. Participants were asked to rate the extent to which each item reflected their feelings and thoughts in their relationships on a 7-point Likert scale (1 = never, 4 = sometimes, 7 = always/continuously). 4 of the items are to apologize/confess (e.g., "I tell my partner that I regret what I did (or did not do)"), 4 of them are to explain/give reason (e.g., "I tell my partner the reasons/reasons for what I did"), 7 of them measure compromising/forgiveness (eg, "I promise to be a better wife in the future") and 5 denial (eg, "I try to minimize/downplay the situation") sub-dimensions.

SECONDARY OUTCOMES:
Burnout Scale Short Form | one day
  The Burnout Scale Short Version consists of 10 items with response options ranging from 1 (Never) to 7 (Always). In the factor analysis study, it was shown that the items were collected in three factors explaining 64.8% of the total variance, but the tool could be evaluated as one-dimensional. It has been observed that those who score high on the scale report more complaints such as chronic fatigue, headaches and backaches than those with low scores, and they have low job satisfaction and low performance expectations. Original Burnout Scale Short Version scores are negatively associated with life satisfaction, general optimism, and job satisfaction. It also showed positive associations with somatic disorder, general work stress, and various specific work stressors.

CONTACTS AND LOCATIONS:
Overall Officials: Berna ERSOY ÖZCAN, Principal Investigator — Sinop University

IPD SHARING:
Plan to Share IPD: No